CLINICAL TRIAL: NCT07018765
Title: The Effect of Mindfulness-Based Stress Reduction Program on Birth Memory and Perception of Traumatic Birth: A Randomized Controlled Trial
Brief Title: Effect of Mindfulness-Based Stress Reduction on Birth Memory and Perception of Traumatic Birth
Acronym: MBSR-BIRTH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kader ATABEY (Other)
Collaborators: Malatya Egitim Ve Arastirma Hastanesi (Other Government)
Responsible Party: Sponsor-Investigator, Kader ATABEY, Assistant Research, Faculty of Health Sciences, Inonu University, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBSR-BIRTH
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Psychological Stress; Mindfulness-Based Stress Reduction; Maternal Health; Traumatic Birth
Keywords: Mindfulness; Postpartum Stress; Maternal Mental Health; Midwifery
MeSH Terms: conditions — Birth Injuries | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial (MBSR vs. control)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR Group (Experimental): Participants in this group will receive an 8-week Mindfulness-Based Stress Reduction (MBSR) program, including weekly 60-90 minute sessions covering mindful breathing, body awareness, emotion regulation, and stress management. The first session will be face-to-face, and subsequent sessions will be delivered online (Zoom).
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Control Group (No Intervention): Participants in this group will receive routine postpartum care and no additional intervention.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — The MBSR program consists of eight weekly sessions, each lasting 60-90 minutes. The first session will be delivered face-to-face in the hospital, and the remaining sessions will be conducted online via Zoom. The program content includes mindful breathing, body scanning, stress management, emotional regulation, and interpersonal mindfulness exercises.
  Arms: MBSR Group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of a Mindfulness-Based Stress Reduction (MBSR) program on birth memory and perception of traumatic birth among women who have undergone vaginal delivery. The study will be conducted between July and October 2025 at Malatya Training and Research Hospital. Participants in the intervention group will attend an 8-week MBSR program, while the control group will receive no intervention. Data will be collected using validated scales before and after the intervention. The primary outcomes are changes in birth memory and traumatic birth perception scores.

DETAILED DESCRIPTION:
This study is a pretest-posttest control group experimental design conducted to determine the effects of a Mindfulness-Based Stress Reduction (MBSR) program on birth memory and the perception of traumatic birth. The population of the study will consist of women who have had a vaginal delivery and received postpartum care at Malatya Training and Research Hospital between July and October 2025. The sample will include 80 women, with 40 in the experimental group and 40 in the control group. The intervention group will participate in an 8-week MBSR program, which includes weekly 60-90 minute sessions-first face-to-face and the rest conducted online. The program content will cover mindful breathing, body awareness, stress and emotion regulation, and interpersonal mindfulness.

Data will be collected using the Mindfulness Scale, the Birth Memory and Recall Scale, and the Traumatic Birth Perception Scale. Pre-test data will be collected during the initial hospital visit, and post-test data will be collected at the end of the 8-week program. No intervention will be applied to the control group. Statistical analyses will include descriptive statistics, independent samples t-tests, and paired samples t-tests. Ethical approval has been applied for and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Women who have undergone a vaginal birth
* Literate and able to understand Turkish
* No diagnosed psychiatric disorder
* Have access to internet and a smart device (for online MBSR sessions)

Exclusion Criteria:

* History of pregnancy loss, stillbirth, or neonatal death
* Complications during postpartum period in mother or newborn
* Incomplete data collection or failure to attend MBSR sessions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in Birth Memory Score | Baseline and 8 weeks post-intervention
  Assessed by the Birth Memory and Recall Scale. Measures the quality and nature of the memory related to the childbirth experience.Assessed by the Birth Memory and Recall Scale (range 6-147). Higher scores indicate more vivid, intense, and emotionally charged birth memories. Items are rated on a 7-point Likert scale. Items 1, 3, and 11 are reverse scored.

SECONDARY OUTCOMES:
Change in Perception of Traumatic Birth | Baseline and 8 weeks post-intervention
  Measured using the Traumatic Birth Perception Scale to evaluate psychological responses and perceived trauma related to childbirth.Measured using the Traumatic Birth Perception Scale (range 0-130). Each item is scored from 0 to 10. Higher scores indicate a higher level of perceived trauma related to childbirth.

OTHER OUTCOMES:
Change in Mindfulness Level | Baseline and 8 weeks post-intervention
  Assessed by the State Mindfulness Scale (range 21-105). Each item is scored from 1 to 5. Higher scores reflect greater mindfulness during the present moment.Assessed by the State Mindfulness Scale (range 21-105). Each item is scored from 1 to 5. Higher scores reflect greater mindfulness during the present moment.

CONTACTS AND LOCATIONS:
Locations (1):
- Malatya Education and Research Hospital, Malatya, Leave Blank, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No